CLINICAL TRIAL: NCT03209648
Title: A Phase 1, Open-Label, Fixed Sequence Study to Investigate the Effect of Itraconazole on the Pharmacokinetics of Debio 1450 in Healthy Subjects
Brief Title: A Study to Investigate the Effect of Itraconazole on the Pharmacokinetics of Debio 1450 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Debio 1450-111; 2017-001352-60 (EudraCT Number)
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Healthy Participants
MeSH Terms: interventions — afabicin; Itraconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Debio 1450 (Experimental): In Treatment Period 1, participants will receive single oral dose of Debio 1450 40 mg on Day 1. In Treatment Period 2, participants will receive itraconazole 200 mg, twice daily (BID) orally, on Day 1, followed by itraconazole 200 mg once daily (QD), on Days 2 to 4, and then single oral dose of Debio 1450 40 mg and itraconazole 200 mg on Day 5, followed by a single oral dose of itraconazole 200 mg on Days 6 and 7.
  Interventions: Drug: Debio 1450; Drug: Itraconazole

INTERVENTIONS:
Drug: Debio 1450 — Debio 1450, 40 mg capsule.
Drug: Itraconazole — Itraconazole, 20 mL of 10 mg/mL solution.

SUMMARY:
Debio 1450 is metabolised mainly by CYP3A4, therefore inhibitors of CYP3A4 have the potential to raise Debio 1450 plasma concentrations. Hence, it is important to determine the effect of CYP3A4 inhibition by itraconazole on the Pharmacokinetics of Debio 1450.

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception.
* Is willing and able to comply with restrictions related to food, drink and medications.
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures.

Exclusion Criteria:

* Has history or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters.
* Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  * the safety or well-being of the participant or study staff.
  * the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding); the analysis of results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Debio 1452 | Days 1 and 5: predose and 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 30, 36, 48, and 60 hours postdose
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUC0-∞) of Debio 1452 | Days 1 and 5: predose and 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 30, 36, 48, and 60 hours postdose
Area Under the Plasma Concentration-time Curve from Time Zero to Time (t) (AUC0-t) of Debio 1452 | Days 1 and 5: predose and 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 30, 36, 48, and 60 hours postdose

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Curve from Time Zero to 12 Hours Postdose (AUC0-12) of Debio 1452, Debio 1450, Debio 1452-M1, and desmethyl Debio 1452 | Days 1 and 5: predose and 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 30, 36, 48, and 60 hours postdose
Time to Reach Maximum Concentration (Tmax) of Debio 1452, Debio 1450, Debio 1452-M1, desmethyl Debio 1452 and Itraconazole | Debio 1450 and its metabolites: Days 1 and 5: predose and 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 30, 36, 48, and 60 hours postdose. Itraconazole: Days 1, 3, and 6: predose, Days 4 and 5: predose, and 0.5, 1, 2, 3, 4, 6, 8, 12 hours postdose
Apparent Plasma Terminal Elimination Half-life (t1/2) of Debio 1452, Debio 1450, Debio 1452-M1, desmethyl Debio 1452 and Itraconazole | Debio 1450 and its metabolites: Days 1 and 5: predose and 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 30, 36, 48, and 60 hours postdose. Itraconazole: Days 1, 3, and 6: predose, Days 4 and 5: predose, and 0.5, 1, 2, 3, 4, 6, 8, 12 hours postdose
Mean Residence Time (MRT) of Debio 1452, Debio 1450, Debio 1452-M1, and desmethyl Debio 1452 | Days 1 and 5: predose and 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 30, 36, 48, and 60 hours postdose
  the mean residence time is the average time the drug stays at the site of action.
Apparent Total Body Clearance of a Drug from the Plasma (CL/F) of Debio 1452 | Days 1 and 5: predose and 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 30, 36, 48, and 60 hours postdose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Apparent Volume of Distribution During the Terminal (lamdaz) Phase (Vz/F) of Debio 1452 | Days 1 and 5: predose and 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 30, 36, 48, and 60 hours postdose
  Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug.
Maximum Observed Plasma Concentration (Cmax) of Debio 1450, Debio 1452-M1, desmethyl Debio 1452 and Itraconazole | Debio 1450 and its metabolites: Days 1 and 5: predose and 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 30, 36, 48, and 60 hours postdose. Itraconazole: Days 1, 3, and 6: predose, Days 4 and 5: predose, and 0.5, 1, 2, 3, 4, 6, 8, 12 hours postdose
Area Under the Plasma Concentration-time Curve from Time Zero to Time (t) (AUC0-t) of Debio 1450, Debio 1452-M1 and desmethyl Debio 1452 | Days 1 and 5: predose and 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 30, 36, 48, and 60 hours postdose
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUC0-infinity) of Debio 1450, Debio 1452-M1 and desmethyl Debio 1452 | Days 1 and 5: predose and 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 30, 36, 48, and 60 hours postdose
Metabolite:Parent Cmax Ratio (for Debio 1452-M1 and desmethyl Debio 1452 only; Debio 1452 as Parent; Based on Molar Data) | Days 1 and 5: predose and 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 30, 36, 48, and 60 hours postdose
Metabolite:Parent AUC ratio (for Debio 1452-M1 and desmethyl Debio 1452 only; Debio 1452 as Parent; Based on Molar Data) | Days 1 and 5: predose and 0.5, 1, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 30, 36, 48, and 60 hours postdose
Area Under the Plasma Concentration-time Curve During a Dosing Interval at Steady State (AUC0-τ) of Itraconazole | Days 1, 3, and 6: predose Days 4 and 5: predose, and 0.5, 1, 2, 3, 4, 6, 8, 12 hours postdose
Measured Concentration at the end of a Dosing Interval at Steady State (Ctrough) of Itraconazole | Days 1, 3, and 6: predose Days 4 and 5: predose, and 0.5, 1, 2, 3, 4, 6, 8, 12 hours postdose
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to Week 7
  An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A Serious Adverse Event (SAE) is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit Ltd., Leeds, United Kingdom